CLINICAL TRIAL: NCT06332027
Title: Accuracy of Hystro-Salpingo-Foam-Sonography (HYFOSY) as Tubal Patency Test in Comparison to Laparoscopy in Infertile Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed, Assistant lecturer Obstetrics and Gynecology Department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-24-03-03MD
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hystro-Salpingo-Foam-Sonography (HYFOSY) — antibiotic prophylaxis oral azithromycin 500 mg per day 3 days the patient lie in dorsal lithotomy cervix visualized by Cusco speculum, cleaned with betadine 7% 6-Fr pediatric Foley's balloon catheter will be introduced into the cervical canal inflated with 2 ml of saline to prevent backflow of contrast through the cervix TV-US probe will be introduced,The foam will be created by mixing 3-4ml of 2% rialocaine gel (lidocaine hydrochloride 2%, Riadh Pharma,Saudi Arabia) with 16-17 ml of saline shaking the mixture between two syringes until a whitish suspension 20ml of lidocaine foam infused into uterine cavity observing the flow in each fallopian tube using greyscale and power Doppler (PD) 2D ultrasound Foam flow over the whole length of the tube fimbrial outflow, or peritoneal spillage of contrast provided evidence of tubal patency Patients observed for15-30 min for any complication or increase in pain Comparison between results and that of laparoscopy in operative list

SUMMARY:
Tubal patency testing is an essential part of female subfertility evaluation . Tubal abnormalities are seen in 30-40% of female subfertility patients . Laparoscopy with chromopertubation is considered to be the gold standard diagnostic procedure .

Laparoscopy is an invasive test, with a risk of intra-abdominal bleeding, visceral damage, and risks related to general anaesthesia.

Traditionally, Hysterosalpingography(HSG) is a less invasive less expensive first-step alternative, which has been used for decades with disadvantages such as radiation exposure, discomfort, or even abdominal pain.

Hysterosalpingo-Contrast Sonography (HyCoSy) was introduced as an alternative using either contrast media or saline. The accuracy of HyCoSy is comparable to that of HSG and LSC being reference standards for tubal patency testing.However, hyperechogenic contrast media such as Echovist_ (Schering AG, Berlin) and SonoVue_ (Bracco, Milan)are either no longer available or not licensed for tubal patency testing.

Hysterosalpingo-Foam Sonography (HyFoSy) was developed as an alternative for contrast HyCoSy and was introduced in 2010 as a first-line office tubal patency test.Foam is used in the HyFoSy technique to visualize the fallopian tubes and is created by rigorously mixing 5mlExEm_-gel (containing hydroxyethyl cellulose and glycerol,IQMedical Ventures BV, Rotterdam, TheNetherlands) with 5ml purified ExEm_-water.

The ExEm_-foam is sufficiently fluid to pass the fallopian tubes and in the mean time sufficiently stable to show echogenicity for at least five minutes, which is an advantage over saline. In a review on safety aspects and side effects of ExEm-gel it was considered to be appropriate and safe for tubal patency testing.

In 2017, HyLiFoSy combined with power Doppler (PD)(HyLiFoSy-PD) technique was described as a possibly less painful and easier to detect on ultrasound alternativeto HyFoSy and HyCoSy, which can be used whenever the contrast media used with both are either unavailable or is relatively expensive Ultrasound-based tubal patency tests include hysterosalpingo-contrast sonography (HyCoSy), hysterosalpingo-foam sonography (HyFoSy), and hysterosalpingo-lidocaine-foam sonography (HyLiFoSy)and have shown a high detection rate of tubal obstruction and good reproducibility with concordances from 83.8 to 100% with HSG, and from 78.1 to96.91% with lap-and-dye test.

In addition, they allow for a single comprehensive assessment of the uterus and the fallopian tubes and it can be performed by the same specialist who indicates it, in the clinician's own office with it consequently being time efficient. Finally, some studies have shown an increase in the rate of post-procedure gestation.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-40
2. Sexually active
3. Infertility or subfertility primary and secondary

Exclusion Criteria:

1. Current pregnancy
2. Heavy menstrual bleeding
3. Peivic inflammatory disease
4. Allergy to lidocaine

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
the accuracy of HyFoSy in the assessment of tubal patency | 1yr
  by comparing it with the reference standard of LDT, using the measures of diagnostic accuracy: sensitivity, specificity,positive predictive value (PPV), negative predictive value (NPV), positive likelihood ration (LR), negative LR, and overall accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fertility problems: assessment and treatment. London: National Institute for Health and Care Excellence (NICE); 2017 Sep. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK554709/ PMID 32134604
- [Background] Exalto N, Emanuel MH. Clinical Aspects of HyFoSy as Tubal Patency Test in Subfertility Workup. Biomed Res Int. 2019 Jul 8;2019:4827376. doi: 10.1155/2019/4827376. eCollection 2019. PMID 31360713
- [Background] Melcer Y, Zilberman Sharon N, Nimrodi M, Pekar-Zlotin M, Gat I, Maymon R. Hysterosalpingo-Foam Sonography for the Diagnosis of Tubal Occlusion: A Systematic Review and Meta-analysis. J Ultrasound Med. 2021 Oct;40(10):2031-2037. doi: 10.1002/jum.15607. Epub 2020 Dec 28. PMID 33368463
- [Background] Piccioni MG, Riganelli L, Filippi V, Fuggetta E, Colagiovanni V, Imperiale L, Caccetta J, Panici PB, Porpora MG. Sonohysterosalpingography: Comparison of foam and saline solution. J Clin Ultrasound. 2017 Feb;45(2):67-71. doi: 10.1002/jcu.22412. Epub 2016 Oct 18. PMID 27753111